CLINICAL TRIAL: NCT05085639
Title: Phase I Study of the Safety, Tolerability and Immunogenicity of GLS-5310 DNA Vaccine Against SARS-CoV-2
Brief Title: GLS-5310 Vaccine in Healthy Volunteers for the Prevention of SARS-CoV-2 (COVID-19)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GeneOne Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CoV2-002
Record Dates: First submitted 2020-12-23; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Healthy
Keywords: Vaccine; DNA
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GLS-5310 1.2 mg (Group 1) (Experimental): GLS-5310 1.2 mg (ID + Gene-Derm) at Day 0 and Week 8
  Interventions: Biological: GLS-5130
- GLS-5310 2.4 mg (Group 2) (Experimental): GLS-5310 1.2 mg (ID + Gene-Derm) + 1.2 mg (IN) at Day 0 and Week 8
  Interventions: Biological: GLS-5130
- GLS-5310 1.2 mg (Group 3) (Experimental): GLS-5310 1.2 mg ID at Day 0 and Week 8
  Interventions: Biological: GLS-5130
- Placebo (Group 4) (Placebo Comparator): Placebo (ID + Gene-Derm) at Day 0 and Week 8
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GLS-5130 — GLS-5310 DNA plasmid vaccine
  Arms: GLS-5310 1.2 mg (Group 1); GLS-5310 1.2 mg (Group 3); GLS-5310 2.4 mg (Group 2)
Biological: Placebo — Placebo
  Arms: Placebo (Group 4)

SUMMARY:
Phase I study of the safety, tolerability and immunogenicity of GLS-5310 DNA vaccine against SARS-CoV-2 (COVID-19)

DETAILED DESCRIPTION:
This Phase I, randomized, placebo-controlled, dose-ranging, single-blind study will assess the safety, tolerability, and immunogenicity of GLS-5310 DNA vaccine administered intradermally (ID) with or without concomitant intranasal (IN) administration of GLS-5310. Vaccine delivered ID will either be performed by Mantoux injection and followed by suction applied to the skin surface using the Gene-Derm device or Mantous injection alone without applied suction. Vaccine delivered IN will be administered using the MAD300 atomizer.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 to 65 years of age
2. Able to provide informed consent
3. Able and willing to comply with study procedures
4. For women of childbearing potential, able and willing to use an approved form of pregnancy prevention during the study
5. Negative test result for the presence of SARS-CoV-2 IgM and IgG antibodies, which indicate recent or prior infection

Exclusion criteria:

1. Persons involved in the care of patients with COVID-19 and health care workers considered, in the opinion of the investigator, to be at increased risk of infection from SARS-CoV-2
2. Persons with symptoms in the past 2 weeks consistent with possible acute SARS-CoV-2 infection to include fever, loss of smell or taste
3. Persons diagnosis of type 2 diabetes mellitus
4. Persons with a diagnosis of chronic kidney disease
5. Persons with a diagnosis of chronic obstructive pulmonary disease (COPD)
6. Persons with a diagnosis of heart conditions to include heart failure, coronary artery disease, prior heart attack, cardiomyopathy
7. Obesity (BMI of 30 kg/m2 or greater)
8. Sickle cell disease
9. Current or former smoker
10. Current or planned pregnancy during the study
11. Currently breastfeeding
12. Current or past participation in a coronavirus (MERS-CoV, SARS-CoV-2) vaccine study, or receipt of a SARS-CoV-2 vaccine that has been approved by the FDA, including vaccines that have received Emergency Use Authorization (EUA)
13. Administration of an investigational agent within 90 days of the 1st dose
14. Administration of a vaccine within 2 weeks prior to the 1st dose
15. Administration of immune globulin within 6 months of enrollment
16. Administration of an anti-TNFα inhibitor such as infliximab, adalimumab, etanercept, or anti-CD20 monoclonal antibody rituximab within 6 months from enrollment
17. Current daily treatment of systemic corticosteroids of 20 mg of prednisone or greater; or the equivalent dose of other systemic corticosteroids
18. Treatment within the four weeks prior to enrollment with any drug intended for the prophylaxis or treatment of COVID-19
19. Any prior treatment with an anti-SARS-CoV-2 monoclonal antibody or immune serum
20. Prior treatment with an anti-IL-6 inhibitor, anti-IL-1 inhibitor, anti-TNF monoclonal antibody, or anti-JAK inhibitor (see Appendix B exclusionary period for specific drugs)
21. History of malignancy
22. History of transplantation (any organ or bone marrow)
23. Current or planned chemotherapy treatment for hematologic or solid tumor during study period
24. History of other congenital or acquired immunodeficiency, excluding those with HIV infection who are taking highly active antiretroviral therapy and who have documentation of undetectable serum viral load
25. History of PCR-confirmed infection with SARS-CoV-2
26. Not willing to allow storage and future use of samples for SARS-CoV-2 related research and who have a CD4 count > 200 cells/µL on two measures at least 3 months apart
27. Prisoner or subjects who are compulsorily detained for treatment of a psychiatric illness
28. Any illness or condition that, in the opinion of the investigator, may affect the safety of the subject or the evaluation of a study endpoint

    Exclusion criteria (ID + IN only):
29. History of chronic rhinosinusitis
30. History of nasal septal defect or deviated nasal septum
31. History of cleft palate
32. History of nasal polyps
33. History of other disorders that, in the opinion of the investigator, may adversely affect administration of intranasal vaccine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 56 weeks post vaccination
  solicited/unsolicited local and systemic AEs
Geometric mean titer (GMT) of antigen specific antibody titers | Through 56 weeks post vaccination
  Endpoint titer of binding antibody in serum

SECONDARY OUTCOMES:
Evaluation of positive response rate of T cell responses induced by GLS-5310 | Through 56 weeks post vaccination
  T-cell response of antigen-specific interferon - gamma (IFN-γ) secretion in PBMC at each timepoint
Geometric mean titer (GMT) of neutralizing antibody titers | Through 56 weeks post vaccination
  Plaque-reduction neutralizing titer(PRNT) in serum at each timepoint

OTHER OUTCOMES:
Determine IgG antibody responses after a single dose of GLS-5310 related to treatment arm | Through 56 weeks post vaccination
  Endpoint titer of binding antibody in serum at each timepoint
Determine IgA antibody responses following vaccination of GLS-5310 related to treatment arm | Through 56 weeks post vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- Puerto Rico (2):
  - Clinical Research Puerto Rico, San Juan, PR
  - University of Puerto Rico, San Juan